CLINICAL TRIAL: NCT04803448
Title: Patient Doctor Lies: When is Privacy Assurance a Bad Thing? A Randomized Clinical Trial
Brief Title: Patient Doctor Lies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Tamara Masters, PhD, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-059
Record Dates: First submitted 2021-03-04; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Patient Lying; Privacy Statements; Risk Statements; Benefit Statements; Patient Lie Detection
Keywords: patient lies; lie detection; privacy; risk; benefits
MeSH Terms: interventions — Privacy; Risk

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned one of 1 intervention statements and then asked health care questions. This is a between subject 6 cell study, the dependent variable is the amount of lying as measured by answer adjustment and biometric mouse-movement under each intervention statement.
Who Masked: Participant
Masking Description: All participants respond to a request to take an online survey about health. Participants are blind to the purpose of the study and do not know what intervention group they are randomly assigned to by the survey software. Participants intervention is numerically coded so during analysis it is not evident what intervention statement the participant saw.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (No Intervention): No statement is provided before asking the health care question. Example: What is your weight in pounds?
- Benefit Statement (Experimental): A statement of benefit will be given (see intervention) after the health question.
  Interventions: Behavioral: Benefit statement
- Risk Statement (Experimental): A statement of risk will be given (see intervention) after the health question.
  Interventions: Behavioral: Risk Statement
- Privacy Statement (Experimental): A statement of privacy will be given (see intervention) after the health question.
  Interventions: Behavioral: Privacy Statement
- Benefit + Privacy statement (Experimental): A statement of benefit and privacy will be given (see intervention) after the health question.
  Interventions: Behavioral: Benefit + Privacy
- Risk + privacy statement (Experimental): A statement of risk and privacy will be given (see intervention) after the health question.
  Interventions: Behavioral: Risk + Privacy

INTERVENTIONS:
Behavioral: Benefit statement — The participant reads this statement after asked one of eight health questions
  1. What is your height in inches?
  2. What is your weight in pounds?
  3. How many days out of the last 2 weeks did you drink alcohol?
  4. How often a month do you use other substance such as marijuana, cocaine, ecstasy, or other drugs
  5. How often a month do you use Rx or non-Rx medications to excessive amounts?
  6. When was the last time you smoked a cigarette?
  7. How many days in the last 2 weeks did you engage in more than 30 min exercise?
  8. How many times did you engage in sexual activity in the last month with another individual? . The statement reads: Accurately answering this will increase the likelihood of a correct diagnosis.
  An example of this with one of the 8 health questions is... What number of days in the last 2 weeks you engaged in >30 minutes of exercise? Accurately answering this will increase the likelihood of a correct diagnosis.
  Arms: Benefit Statement
Behavioral: Risk Statement — The participant reads this statement after being asked one of eight health questions.
  The statement reads: Inaccurately answering this will increase the likelihood of an incorrect diagnosis.
  Arms: Risk Statement
Behavioral: Privacy Statement — The participant reads this statement after being asked one of eight health question for example. "We will not share or sell this personal health information with anyone. We will comply with all HIPPA regulations regarding the protection of your data."
  Arms: Privacy Statement
Behavioral: Benefit + Privacy — The statement reads "Accurately answering this will increase the likelihood of a correct diagnosis. We will not share or sell this personal health information with anyone. We will comply with all HIPPA regulations regarding the protection of your data."
  Arms: Benefit + Privacy statement
Behavioral: Risk + Privacy — The statement reads "Inaccurately answering this will increase the likelihood of an incorrect diagnosis. We will not share or sell this personal health information with anyone. We will comply with all HIPPA regulations regarding the protection of your data."
  Arms: Risk + privacy statement

SUMMARY:
Accurate patient information disclosure is critical to provide optimal treatment. Methods that can detect and then increase the truthfulness of information are relatively unknown.

To investigate the impact of communication about privacy, benefits, and risk on patient truthfulness, the investigators test two new methods to detect patient truthfulness and demonstrate the effects of privacy notices (e.g. HIPPA statements).

Participants include a national online sample randomly assigned to one of six treatment statements that might be typically given before health information was requested. The assigned treatments include one or mix of the following: privacy notice, statement of the benefits of accurate disclosure, and statement of the risks of inaccurate disclosure and control of no statement before being asked typical health questions.

The investigators propose that based on elaboration likelihood model, statements reminding participants of their privacy will increase lying.

The investigators hypothesis the use of a new biometric mouse movement lie detection method and answer adjustment can measure patient lies.

The investigators hypothesis that reminders of the risk of not telling the truth will reduce lying due to risk aversion.

Lastly the investigators hypothesis that statements of benefits of answering truthfully will increase truthfulness.

DETAILED DESCRIPTION:
After agreeing to an IRB-approved modified consent form designed to hide the true purpose of the study to detect lying, all participants will complete the CESD-10 depression scale. This validated measure of depression was used in order to simulate the false pretense of the experiment.

This online survey randomly assigns participating adults to one of six intervention statements after which they are asked eight typical questions about their health. The statements include:

1. control (no stimuli)
2. benefit (statement about the benefits of accurate information disclosure)
3. risk (statement about the risks of inaccurate information disclosure)
4. privacy (a traditional medical privacy notification and seal image)
5. privacy + benefit
6. privacy + risk After this intervention participants are asked to disclose eight items of personal health information, including their weight, height, alcohol intake, illegal drug use, prescription drug abuse, smoking, exercise, and sexual activity. We do not assess these actual numbers. They will be the basis for assessing truthfulness by answer adjustment or biometric mouse-movement.

An example of an intervention benefit statement followed by a health question about weight reads: "What is your weight? Accurately answering this will increase the likelihood of a correct diagnosis." A risk statement reads: "What is your weight? Inaccurately answering this will increase the likelihood of an incorrect diagnosis." A privacy statement read: "What is your weight? We will not share or sell this personal health information with anyone. We will comply with all HIPPA regulations regarding the protection of your data."

The dependent variable - patient truthfulness, will be measured in two ways.

1. First measure of truthfulness will be a biometric mouse-movement measure. As participants answer the health care questions coded programming will measure the mouse-movement arc distance and time to response for biometric lie detection. This measurement is completed when participants move to their response to each health question.
2. Second measure of truthfulness will be the answer adjustment method. Participants will be given a summary of their answers from their health questions in a read-only format and asked to indicate how OVER of UNDERSTATED each initial response was (e.g., "You indicated that your current weight is 185 lbs. How overstated or understated is that value?") on a scale from -5 (understated) to 5 (overstated). The absolute value of their scaled response represents the extent to which participants' initial response deviated from the truth. This the unit of measure to be used in analysis.
3. The answer adjustment values and the mouse tracking results provide a more holistic measure of truthfulness than one alone.

No personal identifiers are collected. Age and gender are collected.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Individuals 18-80 years
* English speaking
* Live in the United States

Exclusion Criteria:

* Participants that do not complete the survey

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-04-19 (Actual)

PRIMARY OUTCOMES:
Patient truthfulness - biometric mouse-movement distance | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  The measure of the distance (mm) the mouse travels to the response.
Patient truthfulness - biometric mouse-movement time | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  The measure of the time (ms) the mouse travels to the response.
Patient truthfulness Weight - answer adjustment from -5 to 5 for each health question | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participants will be given a summary of their answers from their health questions in a read-only format and asked to indicate how over- or understated each initial response was (e.g., "You indicated that your current weight is 185 lbs. How overstated or understated is that value?") on a scale from -5 (understated) to 5 (overstated). The absolute value of their response represents the extent to which participants' initial response deviated from the truth. Participant's actual response to the health questions are NOT an outcome measure but rather how much they adjust their answer on a scale of (-5 to +5).
Patient truthfulness Height - answer adjustment from -5 to 5 for each health question | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participant will be shown a summary of their answer from their health question (What is your height in inches) and then respond to how much they under represented the information (-5) to being accurate (0) to overstated the information (+5). Participant response will be on a sliding scale -5 to +5
Patient truthfulness Drink Alcohol - answer adjustment from -5 to 5 for each health question | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participant will be shown a summary of their answer from their health question (How many days out of the last 2 weeks did you drink alcohol? (1 = 0 time; 6 = 13-14 times)) and then respond to how much they under represented the information (-5) to being accurate (0) to overstated the information (+5). Participant response will be on a sliding scale -5 to +5
Patient truthfulness Drug Activity - answer adjustment from -5 to 5 for each health question | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participant will be shown a summary of their answer from their health question (How often a month do you use other substance such as marijuana, cocaine, ecstasy, or other drugs (1 = never; 6 = all the time)) and then respond to how much they under represented the information (-5) to being accurate (0) to overstated the information (+5). Participant response will be on a sliding scale -5 to +5
Patient truthfulness Prescription Use - answer adjustment from -5 to 5 for each health question | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participant will be shown a summary of their answer from their health question (How often a month do you use Rx or non-Rx medications to excessive amounts? (1 = never; 6 = all the time)) and then respond to how much they under represented the information (-5) to being accurate (0) to overstated the information (+5). Participant response will be on a sliding scale -5 to +5
Patient truthfulness Cigarette Smoking- answer adjustment from -5 to 5 for each health question | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participant will be shown a summary of their answer from their health question (When was the last time you smoked a cigarette? (1 = 6+ weeks ago to 6 = today)) and then respond to how much they under represented the information (-5) to being accurate (0) to overstated the information (+5). Participant response will be on a sliding scale -5 to +5
Patient truthfulness Exercise Activity- answer adjustment from -5 to 5 for each health question | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participant will be shown a summary of their answer from their health question (How many days in the last 2 weeks did you engage in more than 30 min exercise? (1 = 13-14 times; 6 = 0 times)) and then respond to how much they under represented the information (-5) to being accurate (0) to overstated the information (+5). Participant response will be on a sliding scale -5 to +5
Patient truthfulness Sexual Activity - answer adjustment from -5 to 5 for each health question | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participant will be shown a summary of their answer from their health question (How many times did you engage in sexual activity in the last month with another individual? (1 = 0; 6 = 20+ times)) and then respond to how much they under represented the information (-5) to being accurate (0) to overstated the information (+5). Participant response will be on a sliding scale -5 to +5

SECONDARY OUTCOMES:
Gender | The time frame of data collection will be from when the survey is opened by the participant until it is completed and submitted. This will take 10 - 20 minutes.
  Participants will record their gender they identify with - Male or Female

CONTACTS AND LOCATIONS:
Overall Officials: Mark Keith, PhD, Principal Investigator — Brigham Young University
Locations (1):
- Brigham Young University, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: No
The IRB does not allow for sharing of individual participant data

REFERENCES:
- [Background] Levy AG, Scherer AM, Zikmund-Fisher BJ, Larkin K, Barnes GD, Fagerlin A. Prevalence of and Factors Associated With Patient Nondisclosure of Medically Relevant Information to Clinicians. JAMA Netw Open. 2018 Nov 2;1(7):e185293. doi: 10.1001/jamanetworkopen.2018.5293. PMID 30646397
- [Background] Jerrold L. Litigation, legislation, and ethics. When patients lie to their doctors. Am J Orthod Dentofacial Orthop. 2011 Mar;139(3):417-8. doi: 10.1016/j.ajodo.2010.09.004. No abstract available. PMID 21392699
- [Background] Petty RE, Cacioppo JT. The elaboration likelihood model of persuasion. Advances in Experimental Social Psychology. 1986;19:123-205
- [Background] Lowry PB, Moody G, Vance A, Jensen M, Jenkins J, Wells T. Using an elaboration likelihood approach to better understand the persuasiveness of website privacy assurance cues for online consumers. Journal of the American Society for Information Science and Technology. 2012;63(4):755-776
- [Background] Buhrmester M, Kwang T, Gosling SD. Amazon's Mechanical Turk: A New Source of Inexpensive, Yet High-Quality, Data? Perspect Psychol Sci. 2011 Jan;6(1):3-5. doi: 10.1177/1745691610393980. Epub 2011 Feb 3. PMID 26162106
- [Background] Kahneman D, Tversky A. Prospect theory: an analysis of decision under risk. Econometrica. 1979;47(2):263-291
- [Background] Jenkins JL, Proudfoot J, Valacich J, Grimes GM, Nunamaker Jr JF. Sleight of hand: identifying concealed information by monitoring mouse-cursor movements. Journal of the Association for Information Systems. 2019;20(1):1-32
- [Background] Keith MJ, Thompson SC, Hale J, Lowry PB, Greer C. Information disclosure on mobile devices: re-examining privacy calculus with actual user behavior. International Journal of Human-Computer Studies. 2013;71(12):1163-1173
- [Background] DePaulo BM, Kashy DA, Kirkendol SE, Wyer MM, Epstein JA. Lying in everyday life. J Pers Soc Psychol. 1996 May;70(5):979-95. PMID 8656340
- [Background] Argo JJ, White K, Dahl DW. Social comparison theory and deception in the interpersonal exchange of consumption information. Journal of Consumer Research. 2006;33(1):99-108
- [Background] Marchewka A, Jednorog K, Falkiewicz M, Szeszkowski W, Grabowska A, Szatkowska I. Sex, lies and fMRI--gender differences in neural basis of deception. PLoS One. 2012;7(8):e43076. doi: 10.1371/journal.pone.0043076. Epub 2012 Aug 29. PMID 22952631
- See also: Lies patients and doctors tell — https://www.medicareadvantage.com/patient-doctor-lies-survey